CLINICAL TRIAL: NCT01298973
Title: Dispervise Ophthalmic Viscoelastic as an Agent to Ensure Watertight Wound Closure After Clear Corneal Cataract Incisions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Annie Christensen, CRO
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alcon2011-VIS-001
Record Dates: First submitted 2011-01-28; First posted 2011-02-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — chondroitin sulfate, sodium hyaluronate drug combination; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Experimental): One group will receive Saline to irrigate the wound
  Interventions: Drug: Saline
- Viscoat (Experimental): One group will receive Viscoat to close the surgical wound
  Interventions: Drug: Viscoat

INTERVENTIONS:
Drug: Viscoat — One group will receive Viscoat for incision closure
  Arms: Viscoat
Drug: Saline — One group will receive Saline to irrigate the wound
  Arms: Saline

SUMMARY:
The purpose of this study is to look at the ability of Viscoat to ensure proper wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent, complete questionnaires, and likely to complete all visits
* Subject must be male or female, of any race, and at least 21 years old
* Undergoing uncomplicated cataract surgery with clear corneal incisions

Exclusion Criteria:

* Subjects with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course
* Acute or chronic disease or illness that would increase risk or confound study results (e.g., uncontrolled diabetes mellitus, immunocompromised,etc.)
* Uncontrolled systemic disease
* Corneal abnormalities (e.g., stromal, epithelial or endothelial dystrophies)
* Subjects who use concurrent topical or systemic medications that may impair healing, including but not limited to:antimetabolites,isotretinoin (Accutane) within 6 months of treatment, and amiodarone hydrochloride (Cordarone) within 12 months of treatment
* Subjects with a history of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis
* Concurrent participation or participation in the last 30 days in any other clinical trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Ensure watertight, patient wound closure after clear corneal cataract incisions | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Eye Physicians of Central Florida, Maitland, Florida